CLINICAL TRIAL: NCT05951127
Title: Additional Local Consolidative Esophagectomy to Traditional Systemic Therapy for Patients With Oligometastatic Resectable ESCC: A Multi-center, Open-label, Randomized Controlled Tial (LEO)
Brief Title: Additional Consolidative Esophagectomy for the Patients With Oligometastatic Resectable ESCC
Acronym: LEO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC3640
Record Dates: First submitted 2023-03-18; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Esophageal Squamous Cell Carcinoma; Oligometastatic Disease
Keywords: Esophageal Squamous Cell Carcinoma; oligometastatic disease; Esophagectomy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional Local Consolidative Esophagectomy Group (Experimental): The patient in this arm will go on esophagectomy base on tracitional systemic therapy.
  Interventions: Procedure: Esophagectomy
- Traditional Systemic Therapy Group (No Intervention): The patients in this arm will receive traditional therapy, including chemotherapy, immunotherapy, radiotherapy, ect.

INTERVENTIONS:
Procedure: Esophagectomy — Esophagectomy for esophageal cancer and regional lymph nodes dissection.
  Arms: Additional Local Consolidative Esophagectomy Group

SUMMARY:
At present, there are relatively clear treatment guidelines for colorectal cancer with oligometastases, while the treatment mode for resectable esophageal cancer with oligometastases is not clear and there is a lack of research results in this field. The aim of this study is to provide evidence of the optimal therapy model for the local resectable esophageal cancer with oligometastases ESCC patients, by investigating whether 2-year OS of the patients could benefit from additional local consolidative esophagectomy.

DETAILED DESCRIPTION:
This study was designed as a multicenter, open-label, randomized controlled prospective clinical study. The experimental group (group A) received additional esophagectomy after 3-month systemic treatment, and the control group (group B) received only systemic treatment. 2-year OS, 3-year PFS and OS were observed in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed ESCC, and stage was evaluated as cT1-4aN0-3 with oligometastases at initial treatment(According to UICC TNM version 8).

   *Oligonucleotides transfer is defined as: there are 3 or less than 3 lesions in single organ(lung, liver, brain or bone), and could be resected, radiofrequency ablation or radiotherapy in 1 radiation fied; Supraclavicular lymph node metastasis is defined as a distant metastases, celiac axis lymph nodes are considered as regional lymph nodes for the patients with lower 1/3 ESCC; Supraclavicular lymph nodes in patients with upper thoracic and cervical esophageal cancer were defined as regional lymph nodes, while abdominal trunk lymph nodes were considered as distant metastases；
2. No new metastatic lesions were found after more than 3 months of systemic treatment, and primary esophageal cancer lesions and regional lymph nodes can be resected R0;
3. No serious internal disease, KPS score ≥90;
4. The evaluation of various organ functions can tolerate surgery, radiotherapy and other treatments;
5. The following laboratory tests confirmed that bone marrow, liver and kidney function met the requirements for study participation: Hemoglobin ≥9.0g/L; White blood cell count ≥3.5×109/L; Neutrophil absolute value (ANC) ≥1.5×109/L; Platelet count ≥100×109/L; Total bilirubin ≤1.5 times the upper limit of normal value; ALT and AST≤2 times the upper limit of normal value; The international standardized ratio of prothrombin time was less than 1.5 times the upper limit of normal value, and part of the thrombin time was within the normal range; Creatinine ≤1.5 times the upper limit of normal value;
6. Physical state ECOG 0-1;
7. Subject must understand and sign the informed consent form.

Exclusion Criteria

1. Patients with double primary cancer;
2. mental patients;
3. Patients with parotid or salivary gland diseases;
4. Mediastinal lymph nodes could not be thoroughly dissected during radical resection of esophageal cancer; Or the oligometastatic lesions cannot receive local treatment due to location and other reasons;
5. Patients with severe emphysema and pulmonary fibrosis;
6. Active infections requiring medical treatment;
7. Existing or co-existing hemorrhagic disease;
8. Other uncontrollable patients who cannot tolerate chemoradiotherapy or surgery;
9. Patients who cannot be thoroughly cleaned due to previous operations;
10. Pregnant or lactating female patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
2-year OS | Dead time from signing the consent form
  2-year overall survival

SECONDARY OUTCOMES:
3-year OS | Dead time from signing the consent form
  3-year overall survival
3 years PFS | Recurrence time from signing the consent form
  Recurrence of new metastasis from singing the consent form

CONTACTS AND LOCATIONS:
Overall Officials: Yin Li, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing